CLINICAL TRIAL: NCT02150343
Title: A Double-Blind, Randomised, Placebo-Controlled, Multi-Centre Field Study to Assess the Efficacy and Safety of HDM-SPIRE in Subjects With a History of House Dust Mite-Induced Rhinoconjunctivitis
Brief Title: Phase II HDM-SPIRE Safety and Efficacy Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TH005
Record Dates: First submitted 2014-05-27; First posted 2014-05-29 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Rhinoconjunctivitis
Keywords: Cat allergy; Rhinoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HMD-SPIRE Treatment 1 (Experimental): 4 x 12 nmol HDM-SPIRE followed by 4 x placebo 4 weeks apart
  Interventions: Drug: HDM-SPIRE; Drug: Placebo
- HDM-SPIRE Treatment 2 (Experimental): 4 x 12 nmol HDM-SPIRE 4 weeks apart followed by a second course of 4 x 12 nmol HDM-SPIRE 4 weeks apart
  Interventions: Drug: HDM-SPIRE
- HDM-SPIRE Treatment 3 (Experimental): 4 x 20 nmol HDM-SPIRE followed by 4 x placebo 4 weeks apart
  Interventions: Drug: HDM-SPIRE; Drug: Placebo
- Placebo (Placebo Comparator): 8 x placebo 4 weeks apart
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HDM-SPIRE — 1 dose every 4 weeks
  Arms: HDM-SPIRE Treatment 2; HDM-SPIRE Treatment 3; HMD-SPIRE Treatment 1
Drug: Placebo — 1 dose every 4 weeks
  Arms: HDM-SPIRE Treatment 3; HMD-SPIRE Treatment 1; Placebo

SUMMARY:
The purpose of this study is to compare the treatment effect of three treatment regimens of HDM-SPIRE vs placebo and to evaluates the treatment effect of HDM-SPIRE on symptoms, rescue medication usage, Quality of Life and Sleep Quality

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years.
* Moderate to severe rhinoconjunctivitis on exposure to HDM for at least 1 years.
* Mean TRSS ≥10
* Positive skin prick test to Der p and Der f.
* Dep p and Der f specific IgE ≥0.7 kU/L

Exclusion Criteria:

* Diagnosis of asthma requiring Global Initiative for Asthma (GINA) Step 3 (www.ginasthma.org)or higher treatment
* FEV1 <80% of predicted.
* Clinically significant confounding symptoms of allergy to seasonal allergens during the final evaluation period.
* Significant symptoms of another clinically relevant illness that is likely to affect scoring of rhinoconjunctivitis symptoms.
* Clinically relevant abnormalities detected on physical examination.
* History of severe drug allergy, severe angioedema or anaphylactic reaction to food.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2014-09; Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (98):
- United States (56):
  - Birmingham, Alabama
  - Huntington Beach, California
  - Long Beach, California
  - Mission Viejo, California
  - Napa, California
  - Orange, California
  - Redwood City, California
  - Rolling Hills Estates, California
  - Roseville, California
  - San Diego, California
  - Walnut Creek, California
  - Waterbury, Connecticut
  - Tallahassee, Florida
  - Tampa, Florida
  - Stockbridge, Georgia
  - Normal, Illinois
  - Shiloh, Illinois
  - Evansville, Indiana
  - Iowa City, Iowa
  - Owensboro, Kentucky
  - Bangor, Maine
  - Bethesda, Maryland
  - Gaithersburg, Maryland
  - Brockton, Massachusetts
  - Minneapolis, Minnesota
  - Plymouth, Minnesota
  - St Louis, Missouri
  - Bellevue, Nebraska
  - Ocean City, New Jersey
  - Teaneck, New Jersey
  - Verona, New Jersey
  - Rochester, New York
  - Rockville Centre, New York
  - Asheville, North Carolina
  - High Point, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Bethlehem, Pennsylvania
  - Blue Bell, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Dallas, Texas
  - Kerrville, Texas
  - Plano, Texas
  - San Antonio, Texas
  - South Burlington, Vermont
  - Henrico, Virginia
  - Bellingham, Washington
  - Seattle, Washington
  - Vancouver, Washington
  - Greenfield, Wisconsin
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (10):
  - Hamilton, Ontario
  - London, Ontario
  - Niagara, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saint Romuald, Quebec
  - Trois-Rivières, Quebec
- France (4):
  - Reims, Marne
  - Gironde, Pessac
  - Bas Rhin, Strasbourg
  - Meurthe-et-Moselle, Vandoeuvre Les Nancy
- Germany (6):
  - Heidelberg, Baden-Wurttemberg
  - Essen, North Rhine-Westphalia
  - Goch, North Rhine-Westphalia
  - Dresden, Saxony
  - Berlin
  - Hamburg
- Italy (7):
  - Ancona, Torrette Di Ancona
  - Genova
  - Milan
  - Parma
  - Pavia
  - Roma
  - Siena
- Netherlands (3):
  - Almere Stad
  - Amsterdam
  - Beek
- South Africa (4):
  - Durban, KwaZulu-Natal
  - eMkhomazi, KwaZulu-Natal
  - Ottawa, KwaZulu-Natal
  - Cape Town, Western Cape
- Spain (8):
  - Sabadell, Barcelona
  - Santander, Cantabria
  - Girona, Catalonia
  - Donostia / San Sebastian, Guipuzcoa
  - Pamplona, Navarre
  - Bilbao, Vizcaya
  - Barcelona
  - Seville

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 715 participants were randomised on to the study through the IRT. However, one participant was inadvertently randomised before eligibility had been confirmed by the PI, and was withdrawn due to a finding of inspiration/expiration wheeze before receiving any study medication. Therefore results refer to 714 participants throughout.
Groups:
- HDM-SPIRE 12 Nmol (4 Administrations): 12 nmol given at 4 weekly intervals (4 administrations)
- HDM-SPIRE 20 Nmol: 20 nmol given at 4 weekly intervals (4 administrations)
- HDM-SPIRE 12 Nmol (8 Administrations): 20 nmol given at 4 weekly intervals (8 administrations)
- HDM-SPIRE Placebo: 8 administrations at 4 weekly intervals
Period: Overall Study
Arm/Group | HDM-SPIRE 12 Nmol (4 Administrations) | HDM-SPIRE 20 Nmol | HDM-SPIRE 12 Nmol (8 Administrations) | HDM-SPIRE Placebo
Started | 180 | 178 | 178 | 178
Completed | 159 | 158 | 166 | 168
Not Completed | 21 | 20 | 12 | 10
Not completed — Adverse Event | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 13 | 10 | 9 | 4
Not completed — Lost to Follow-up | 4 | 4 | 2 | 3
Not completed — Other | 2 | 6 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HDM-SPIRE 12 Nmol (4 Administrations) | HDM-SPIRE 20 Nmol | HDM-SPIRE 12 Nmol (8 Administrations) | HDM-SPIRE Placebo | Total
Number analyzed (Participants) | 180 | 178 | 178 | 178 | 714
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (11.53) | 38.3 (12.40) | 35.5 (11.61) | 36.8 (12.84) | 36.8 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 109 | 120 | 117 | 453
  Male | 73 | 69 | 58 | 61 | 261
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 7 | 12 | 3 | 10 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 22 | 21 | 23 | 13 | 79
  White | 142 | 133 | 144 | 136 | 555
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 12 | 7 | 19 | 46

OUTCOME MEASURES:

1. Primary Outcome: Combined Score of Symptoms and Allergy Medication
Description: The primary endpoint was mean Combined Score (CS) over a 3 week period (50-52 weeks after randomisation) in the HDM-SPIRE treatment groups compared with the mean CS in the placebo group. A higher score indicated more severe symptoms or greater use of allergy rescue medication and thus a low score indicated a better outcome.
  CS = Total Rhinoconjunctivitis Symptom Score (TRSS) + Rescue Medication Score (RMS). Eight symptoms are defined in the TRSS, 4 nasal symptoms: runny nose, sneezing, blocked nose and itchy nose and 4 non-nasal symptoms: itchy eyes; watery eyes; red eyes, and sore eyes. Each symptom was rated in severity on a score of 0-3 (0=absent, 3=severe); TRSS was divided by the number of symptoms (8) to provide an average score per symptom of 0-3.
  The RMS score ranged from 0 (no allergy rescue medication use per day) to 3 (at least one dose of systemic corticosteroid per day). The RMS score was not additive, and therefore the maximum RMS was 3 and the maximum CS was 6.
Time Frame: Weeks 50 to 52 after randomisation
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HDM-SPIRE 12 Nmol (4 Administrations) | HDM-SPIRE 20 Nmol | HDM-SPIRE 12 Nmol (8 Administrations) | HDM-SPIRE Placebo
Number analyzed (Participants) | 160 | 159 | 165 | 168
units on a scale | 1.69 (0.089) | 1.51 (0.089) | 1.40 (0.086) | 1.56 (0.087)

2. Secondary Outcome: Mean RQLQ Score in HDM-SPIRE Treatment Groups Compared With Placebo
Description: The RQLQ (Rhinoconjunctivitis Quality of Life Questionnaire) was completed by subjects at the end of the study (50-52 weeks after randomisation).
  RQLQ is a validated method of assessing quality of life and has 28 questions in seven domains (activity limitation, sleep problems, nasal symptoms, eye symptoms, non-nasal/eye symptoms, practical problems and emotional function). Subjects recalled how their rhinoconjunctivitis had been during the last week and responded to each question on a seven-point scale (0 = no impairment, 6 = maximum impairment). Questions were equally weighted, and the RQLQ score was the mean of the 28 questions and could range from zero to six.
  A higher score indicated greater impact on quality of life and thus a low score indicated a better outcome.
Time Frame: Weeks 50 to 52 after randomisation
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HDM-SPIRE 12 Nmol (4 Administrations) | HDM-SPIRE 20 Nmol | HDM-SPIRE 12 Nmol (8 Administrations) | HDM-SPIRE Placebo
Number analyzed (Participants) | 160 | 158 | 166 | 167
units on a scale | 2.02 (0.098) | 1.76 (0.098) | 1.72 (0.095) | 1.89 (0.095)

3. Secondary Outcome: Participants Assessment of Change in Rhinoconjunctivitis Symptoms Measured by Rating Overall Symptoms at the End of the Study Relative to Baseline
Description: A Global Impression of Change in Rhinoconjunctivitis Symptoms assessment was completed by subjects at the final follow-up visit. Subjects rated their overall allergy symptoms at the end of the study relative to baseline on a seven-point scale as follows:0. very much better; 1. moderately better; 2. a little better; 3. unchanged; 4. a little worse; 5. moderately worse; 6. very much worse.
  For reporting the individual categories were grouped as follows: moderately or very much better; any improvement; no change and any worsening. Subjects could therefore be reported in more than group and the total number reported does not match the overall number of participants analysed.
Time Frame: Weeks 50 to 52 after randomisation
Population: The overall number of participants analysed represents the number of subjects that completed the assessment, not all subjects that completed the study (651) completed the Clinical Global Impression of Change (633).
Measure: Count of Participants; unit: Participants
Arm/Group | HDM-SPIRE 12 Nmol (4 Administrations) | HDM-SPIRE 20 Nmol | HDM-SPIRE 12 Nmol (8 Administrations) | HDM-SPIRE Placebo
Number analyzed (Participants) | 159 | 156 | 158 | 160
Participants
  Moderately or very much better | 55 | 70 | 61 | 64
  Any improvement | 101 | 109 | 103 | 109
  No Change | 45 | 41 | 48 | 43
  Any worsening | 13 | 6 | 7 | 8

4. Secondary Outcome: Mean TRSS in HDM-SPIRE Treatment Groups Compared With Placebo
Description: Mean Total Rhinoconjunctivitis Symptom Score (TRSS) in HDM-SPIRE treatment groups compared with placebo.
  Eight symptoms are defined in the TRSS, 4 nasal symptoms: runny nose, sneezing; blocked nose, and itchy nose and 4 non-nasal symptoms: itchy eyes; watery eyes; red eyes, and sore eyes. Each symptom was rated in severity on a score of 0-3 (0. absent; 1. mild, barely noticeable; 2. moderate, annoying/troublesome; 3. severe, very annoying/very troublesome), therefore TRSS could range from 0 to 24. Higher TRSS reflected more severe symptom scores. Symptoms were scored daily for a period of approximately 3 weeks, 50-52 weeks after randomisation.
Time Frame: Weeks 50 to 52 after randomisation
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HDM-SPIRE 12 Nmol (4 Administrations) | HDM-SPIRE 20 Nmol | HDM-SPIRE 12 Nmol (8 Administrations) | HDM-SPIRE Placebo
Number analyzed (Participants) | 160 | 159 | 165 | 168
units on a scale | 8.96 (0.468) | 8.03 (0.467) | 7.97 (0.451) | 8.16 (0.455)

5. Secondary Outcome: Mean Non-nasal Score in HDM-SPIRE Treatment Group Compared With Placebo
Description: Mean daily Total Non-nasal Symptom Score (TNNSS) in HDM-SPIRE treatment groups compared to placebo. TNNSS was the sum of all the non-nasal symptom scores (itchy eyes; watery eyes; red eyes; sore eyes) and could range from 0 to 12. Higher TNNSS reflected more severe symptoms.
  Subjects rated the severity of each symptom over the last 24 hours as follows: 0. absent; 1. mild, barely noticeable; 2. moderate, annoying/troublesome; 3. severe, very annoying/very troublesome. Symptoms were scored daily for a period of approximately 3 weeks, 50-52 weeks after randomisation.
Time Frame: Weeks 50 to 52 after randomisation
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HDM-SPIRE 12 Nmol (4 Administrations) | HDM-SPIRE 20 Nmol | HDM-SPIRE 12 Nmol (8 Administrations) | HDM-SPIRE Placebo
Number analyzed (Participants) | 160 | 159 | 165 | 168
units on a scale | 3.99 (0.242) | 3.64 (0.242) | 3.53 (0.233) | 3.73 (0.235)

6. Secondary Outcome: Mean Nasal Score in HDM-SPIRE Treatment Group Compared With Placebo
Description: TNSS (Total nasal symptom score) was the sum of all the nasal symptom scores (runny nose; sneezing; blocked nose; itchy nose) and could range from 0 to 12. Higher TNSS reflected more severe symptoms.
  Subjects rated the severity of each symptom over the last 24 hours as follows: 0. absent; 1. mild, barely noticeable; 2. moderate, annoying/troublesome; 3. severe, very annoying/very troublesome. Symptoms were scored daily for a period of approximately 3 weeks, 50-52 weeks after randomisation.
Time Frame: Weeks 50 to 52 after randomisation
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HDM-SPIRE 12 Nmol (4 Administrations) | HDM-SPIRE 20 Nmol | HDM-SPIRE 12 Nmol (8 Administrations) | HDM-SPIRE Placebo
Number analyzed (Participants) | 160 | 159 | 165 | 168
units on a scale | 4.99 (0.244) | 4.40 (0.243) | 4.45 (0.235) | 4.44 (0.237)

7. Secondary Outcome: Mean RMS in HDM-SPIRE Treatment Group Compared With Placebo
Description: Mean RMS (Rescue medication score) in HDM-SPIRE treatment groups compared with placebo groups.
  The use of rhinoconjunctivitis rescue medications was recorded by the subject on a daily basis just before bedtime for approximately 21 days, 50-52 weeks after randomisation and was scored based on a previously published system as follows: 0 = no allergy rescue medication used per day; 0.5 = at least one dose of antihistamine eye drops used per day; 1 = at least one dose of oral antihistamine used per day; 2 = at least one dose of intranasal corticosteroid used per day; 3 = at least one dose of systemic corticosteroid used per day. The score was according to the highest level of rescue medication used and was not additive.
Time Frame: Weeks 50 to 52 after randomisation
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HDM-SPIRE 12 Nmol (4 Administrations) | HDM-SPIRE 20 Nmol | HDM-SPIRE 12 Nmol (8 Administrations) | HDM-SPIRE Placebo
Number analyzed (Participants) | 160 | 159 | 165 | 168
units on a scale | 0.57 (0.048) | 0.51 (0.048) | 0.41 (0.047) | 0.55 (0.047)

8. Secondary Outcome: Number of Days With no Rescue Medication Use in HDM-SPIRE Treatment Group Compared With Placebo
Description: The number of well days, i.e., days with no moderately or severely annoying symptoms and with no rescue medication used was calculated for all subjects over a period of approximately 21 days, 50-52 weeks after randomisation.
Time Frame: Weeks 50 to 52 after randomisation
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | HDM-SPIRE 12 Nmol (4 Administrations) | HDM-SPIRE 20 Nmol | HDM-SPIRE 12 Nmol (8 Administrations) | HDM-SPIRE Placebo
Number analyzed (Participants) | 160 | 159 | 165 | 168
Days | 25.9 (2.90) | 33.5 (2.89) | 33.9 (2.80) | 31.1 (2.812)

ADVERSE EVENTS:
Time Frame: Upto 52 weeks after randomisation
Arm/Group | HDM-SPIRE 12 Nmol (4 Administrations) | HDM-SPIRE 20 Nmol | HDM-SPIRE 12 Nmol (8 Administrations) | HDM-SPIRE Placebo
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/178 | 0/178 | 0/178
Serious Adverse Events (participants affected / at risk) | 6/180 | 4/178 | 4/178 | 3/178
Other Adverse Events (participants affected / at risk) | 120/180 | 110/178 | 140/178 | 124/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDM-SPIRE 12 Nmol (4 Administrations) (N=180) | HDM-SPIRE 20 Nmol (N=178) | HDM-SPIRE 12 Nmol (8 Administrations) (N=178) | HDM-SPIRE Placebo (N=178)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedual haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDM-SPIRE 12 Nmol (4 Administrations) (N=180) | HDM-SPIRE 20 Nmol (N=178) | HDM-SPIRE 12 Nmol (8 Administrations) (N=178) | HDM-SPIRE Placebo (N=178)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 4 (4) | 8 (9) | 9 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2) | 14 (14) | 6 (9)
Headache (Nervous system disorders) | 10 (26) | 11 (30) | 13 (28) | 12 (16)
Nasopharyngitis (Infections and infestations) | 37 (59) | 32 (54) | 38 (54) | 41 (58)
Upper respiratory tract infection (Infections and infestations) | 22 (27) | 24 (32) | 21 (32) | 20 (26)
Sinusitis (Infections and infestations) | 13 (16) | 14 (15) | 15 (15) | 12 (16)
Influenza (Infections and infestations) | 7 (7) | 12 (15) | 15 (15) | 11 (12)
Urinary tract infection (Infections and infestations) | 5 (6) | 7 (7) | 10 (14) | 6 (9)
Bronchitis (Infections and infestations) | 9 (9) | 4 (4) | 6 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Wording included in the clinical protocol - The Investigator and Circassia will normally prepare a manuscript together. To avoid disclosures that may affect the proprietary rights of the Sponsor, the Investigator agrees to allow Circassia the opportunity to review all manuscripts and abstracts 60 days prior to submission for publication. Circassia reserves the right to include the report of this study in any regulatory documentation or submission or in any informational materials.

DOCUMENTS (2):
  • Study Protocol (2015-04-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT02150343/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT02150343/SAP_001.pdf